CLINICAL TRIAL: NCT05381532
Title: Menstrual-phase-dependent Differences in Response to Sleep Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Melissa A. St. Hilaire, Ph.D, Associate Biostatistician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021P002586; R01HL162102 (NIH)
Record Dates: First submitted 2022-04-27; First posted 2022-05-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Sleep Deprivation
Keywords: Sleep Restriction; Women's Health
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants may not know to which study arm they are assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Chronic variable sleep deficiency - follicular phase (Experimental): This will be the first of four arms of controlled sleep manipulation. Participants randomized to this arm will be studied on a chronic variable sleep deficiency schedule during the follicular phase of their menstrual cycle. The exact sleep schedule is not provided in order to keep participants blinded to sleep conditions.
  Interventions: Behavioral: Controlled sleep
- Chronic variable sleep deficiency - luteal phase (Experimental): This will be the second of four arms of controlled sleep manipulation. Participants randomized to this arm will be studied on a chronic variable sleep deficiency schedule during the luteal phase of their menstrual cycle. The exact sleep schedule is not provided in order to keep participants blinded to sleep conditions.
  Interventions: Behavioral: Controlled sleep
- Control sleep - follicular phase (Experimental): This will be the third of four arms of controlled sleep manipulation. Participants randomized to this arm will be studied on a control sleep schedule during the follicular phase of their menstrual cycle. The exact sleep schedule is not provided in order to keep participants blinded to sleep conditions.
  Interventions: Behavioral: Controlled sleep
- Control sleep - luteal phase (Experimental): This will be the fourth of four arms of controlled sleep manipulation. Participants randomized to this arm will be studied on a control sleep schedule during the luteal phase of their menstrual cycle. The exact sleep schedule is not provided in order to keep participants blinded to sleep conditions.
  Interventions: Behavioral: Controlled sleep

INTERVENTIONS:
Behavioral: Controlled sleep — Duration and timing of sleep will be assigned and monitored in a controlled laboratory environment.

SUMMARY:
This study is designed to assess how healthy premenopausal women respond to different patterns of sleep loss at different times in the menstrual cycle.

DETAILED DESCRIPTION:
During a 1.5-week inpatient laboratory protocol, participants will undergo one of two parallel sleep conditions during either the follicular or luteal phase of the menstrual cycle (4 study arms total). Subjects will be randomly assigned to each study arm. During their time in the laboratory, biological samples (e.g., blood) will be collected for assessment of sex steroid hormones and other analyses. Sleep quantity and quality will be monitored and responses on neurobehavioral tests and surveys will be monitored for differences across conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-35 years old
* Regular menstrual cycle between 26-35 days in duration
* Not using any form of hormonal contraception for at least the prior 3 months
* Regular sleep patterns (7-9 hours/night)
* Not taking any medications or supplements
* Weight >110 lb
* BMI between 18.5 and 29.5 kg/m2

Exclusion Criteria:

* Primary sleep disorder
* History of shift work
* Transmeridian travel in the previous 3 months
* Presence of acute or chronic disease, including but not limited to: diabetes, metabolic disorders, psychiatric illness, reproductive disorders
* Current pregnancy, < 6 months postpartum, and/or breastfeeding
* Blood donation in the past 8 weeks
* Extreme morning or evening chronotype

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PVT mean reaction time | The PVT will be administered at frequent intervals over 11 days in a sleep laboratory. Subjects will be in a time-free environment, and not told the sampling frequency.
  The mean reaction time will be calculated across each Psychomotor Vigilance Task (PVT) session. A linear mixed model analysis will be conducted to compare PVT mean reaction time at each time point (multiple points across the study) across all 4 study arms.
PVT lapses in attention | The PVT will be administered at frequent intervals over 11 days in a sleep laboratory. Subjects will be in a time-free environment, and not told the sampling frequency.
  The number of lapses in attention will be counted across each Psychomotor Vigilance Task (PVT) session. A linear mixed model analysis will be conducted to compare PVT lapses in attention at each time point (multiple points across the study) across all 4 study arms.
KSS score | The KSS will be administered at frequent intervals over 11 days in a sleep laboratory. Subjects will be in a time-free environment, and not told the sampling frequency.
  The Karolinska Sleepiness Score (KSS) measures level of sleepiness on a 9-point Likert scale with 1 = Extremely Alert and 9 = Extremely Sleepy. A linear mixed model analysis will be conducted to compare KSS score at each time point (multiple points across the study) across all 4 study arms.
P4/E2 ratio | Biological samples will be collected at frequent intervals over 11 days in a sleep laboratory. Subjects will be in a time-free environment, and not told the sampling frequency.
  The ratio of progesterone (P4) and estradiol (E2) in each sample will be calculated as (P4 ng/ml x 1000)/E2 pg/ml. A linear mixed model analysis will be conducted to compare the P4/E2 ratio at each time point (multiple points across the study) across all 4 study arms.
Core body temperature | Core body temperature will be collected at frequent intervals over 11 days in a sleep laboratory. Subjects will be in a time-free environment, and not told the sampling frequency.
  Core body temperature is measured via rectal thermistor. A linear mixed model analysis will be conducted to compare the core body temperature at each time point (multiple points across the study) across all 4 study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A St. Hilaire, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data that form the basis of a peer-reviewed manuscript will be made available after publication.
Supporting Information: ICF
Time Frame: Release of data forming the basis of a peer-reviewed manuscript will be made available after publication. Release will be consistent with Institutional Review Board, journal, and federal requirements.
Access Criteria: Access may be controlled, e.g., in accordance with the National Institutes of Health.